CLINICAL TRIAL: NCT04137991
Title: Nol-Index Guided Remifentanil Analgesia Versus Standard Analgesia During Moderate-to-High Risk Cardiovascular Surgery: a Randomized Controlled Trial
Brief Title: Nol-Index Guided Remifentanil Analgesia Versus Standard Analgesia During Moderate-to-High Risk Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2019/427
Record Dates: First submitted 2019-10-08; First posted 2019-10-24 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Nociceptive Pain; Goal-directed Therapy; Hemodynamic Instability; Nol-Index; Remifentanil; Cardiac Surgery; Vascular Surgery; General Anesthesia
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nol-Guided Analgesia Group (Experimental): In the Nol-Guided Analgesia Group remifentanil effect site concentration will be adapted to maintain the NOL-index between 10 and 25 throughout the anesthetic.
  Interventions: Device: Nol-Index guided analgesia
- Standard Analgesia Group (Active Comparator): Remifentanil titration in the Standard Analgesia Group will be left at the anesthesiologists discretion (i.e., guided by heart rate, blood pressure, and experience).
  Interventions: Other: Standard Analgesia

INTERVENTIONS:
Device: Nol-Index guided analgesia — Monitor that indicates the level of nociception-antinociception balance
  Arms: Nol-Guided Analgesia Group
Other: Standard Analgesia — Administration of remifentanil based guided by heart rate, blood pressure, and experience
  Arms: Standard Analgesia Group

SUMMARY:
This study will investigate the potential of guiding remifentanil analgesia during cardiac and vascular surgery in moderate to high risk patients requiring general anesthesia.

DETAILED DESCRIPTION:
Justification:

Moderate-to-high risk cardiovascular surgery is associated with perioperative morbidity and mortality. These patients undergo general anesthesia and often require tight blood pressure control (e.g., using norepinephrine titration) to avoid the complications associated with hypotension and reduced cardiac output. Standard analgesia opioid titration to control nociception (i.e., the patient's unconscious response to noxious stimuli) is based on the anesthesiologist's experience and variations in the patient's heart rate and blood pressure. This causes anesthesiologists to often give too much analgesic, which can lead to inhibition of the sympathetic autonomic nervous system, hypotension, and associated side effects. A recently developed nociception monitor, the PMD-200 (Medasense, Israel), is capable of measuring the patient's level of nociception-antinociception balance and can guide opioid administration. This monitor may allow anesthesiologists to administer only the required amount of opioid, which may lead to better hemodynamic stability and better postoperative outcome.

Objectives:

The goal of this study is to determine if titrating analgesia using the Nol-Index, when compared to standard care, leads to decreased infused remifentanil, decreased norepinephrine, increased cardiac output, more stable blood pressure control, and decreased postoperative complications in moderate-to-high risk patients undergoing cardiac or vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-high risk cardiac or vascular surgery
* ASA 2-4

Exclusion Criteria:

* chronic arrhythmia (e.g. atrial fibrillation)
* aortic insufficiency
* pacemaker
* implanted defibrillator
* valve surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Remifentanil requirement | 2 to 8 hours
  µg/kg/hour required during general anesthesia

SECONDARY OUTCOMES:
Norepinephrine requirement | 2 to 8 hours
  µg/kg/hour required during general anesthesia
propofol requirement | 2 to 8 hours
  mg/kg/hour required during general anesthesia
nicardipine requirement | 2 to 8 hours
  mg/kg/hour required during general anesthesia
esmolol requirement | 2 to 8 hours
  mg/kg/hour required during general anesthesia
Intraoperative hemodynamic instability | 2 to 8 hours
  Occurence of hypotension, hypertension, bradycardia or tachycardia
Number of patients with 28 day composite and individual adverse outcomes | 28 days
  renal failure, cardiac ischemia, ileus, stroke, new onset arrhythmia, etc
Heart Rate | 2 to 8 hours
  Heart rate during anesthesia
Systolic Blood Pressure | 2 to 8 hours
  systolic blood pressure during anesthesia
Diastolic Blood Pressure | 2 to 8 hours
  diastolic blood pressure during anesthesia
Mean Blood Pressure | 2 to 8 hours
  mean blood pressure during anesthesia
Cardiac Output | 2 to 8 hours
  cardiac output during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Anesthesia Department, Erasme Hospital, Brussels, Belgium